CLINICAL TRIAL: NCT06552767
Title: Thrombosis and Inflammation in Vessels Initiative (TIVI)
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001781; 001781-H
Record Dates: First submitted 2024-08-07; First posted 2024-08-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Cardiovascular Diseases; Vascular Diseases
Keywords: Vascular
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected Participants and Relatives: Participants with relevant immune, inflammation, thrombotic and/or vascular diseases and their relatives
- Healthy Volunteers: Healthy volunteers

SUMMARY:
Background:

Diseases related to the immune system, blood clots, and blood vessels can affect every part of the body. These diseases are now known to be interrelated: People who have strokes, blood clots in their legs, or autoimmune disease, for example, are at greater risk of complications in the heart, brain, and other organs. Researchers want to learn more about how these diseases start, how they change over time, and how they affect different organs.

Objective:

To learn more about how inflammation and diseases of the blood vessels start and how they change over time.

Eligibility:

People aged 5 years and older with a disease related to blood clots, the immune system, or blood vessels. Healthy relatives of people with these diseases and unrelated healthy volunteers are also needed.

Design:

Participants will have a baseline visit: They will provide a medical history, physical exam and blood test. All other tests and procedures are optional; these may be spread over more than 1 day:

Tests of heart and lung function.

Fill in a family tree form.

Imaging scans

Treadmill or bike stress tests and a 6-minute walk test.

Tests of blood pressure and the flow of blood through vessels.

Photos of the face and body.

Eye exams, with photos taken of the retina.

Saliva and urine samples.

Biopsies (tissues samples) of the skin and fat.

Tests of thinking and mental function.

Evaluations by other medical specialists.

Participants may opt to return for repeat testing for up to 90 months (7.5 years).

Some visits may be done by telehealth.

DETAILED DESCRIPTION:
Study Description:

Thrombotic vascular disorders remain the leading cause of morbidity and mortality in the United States. The proximate determinants of thrombosis, arterial, venous, and lymphatic vascular disorders and their treatments remains incompletely understood. In pursuit of improved vascular health, this disease discovery protocol will facilitate rapid initiation of new clinical and molecular phenotype-specific investigations to collect data and biospecimens on affected individuals, family members, and unrelated healthy controls. The data collected in this protocol will inform the design of future disease-specific investigational protocols.

Objectives:

Primary Objective:

To study the pathogenesis of patients affected with thrombotic, immune, vascular, and cardiovascular conditions including clinical, radiographic, immunological and genetic characteristics of the disease.

Secondary Objectives:

* To develop long-term clinical and laboratory outcome parameters of organ involvement in patients with thrombotic, inflammatory, vascular and cardiovascular diseases
* Evaluation of blood, body fluid, and tissue biomarkers during disease flares and quiescence.
* To develop disease activity indices for vascular disease that incorporate clinical, laboratory, and imaging data.
* Screening for other NHLBI clinical studies
* To evaluate patients referred for suspected vascular disease and provide additional opinions for diagnosis and management recommendations

Endpoints:

This is a disease discovery protocol and there are no specific endpoints associated with this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Age >= 5 years at the time of consent
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document

In addition, the following cohort-specific inclusion criteria apply:

Affected Subjects:

-Known or possible thrombotic, immune, or vascular disorder after review of the subject s medical records and/or discussion of medical history

Relatives of Affected Subjects:

-Being a relative of an affected subject

Unrelated Healthy Controls:

-In good general health as evidenced by medical history

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

-Any condition that in the opinion of the Investigator would warrant exclusion

Unrelated Healthy Controls:

* Unrelated healthy volunteers who decline to have blood drawn and/or tissue studies or who do not consent to have samples stored for future research
* Cognitively impaired individuals

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with relevant immune, inflammation, thrombotic and/or vascular diseases and their relatives Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2034-01-30 (Estimated); Study Completion 2034-01-30 (Estimated)

PRIMARY OUTCOMES:
This is a disease discovery protocol and there are no specific endpoints associated with this protocol. | Study End

CONTACTS AND LOCATIONS:
Overall Officials: Yogendra Kanthi, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from IPD or aggregated data may be shared in publications for scientific data reporting and interpretation.
Supporting Information: Study Protocol, ICF
Time Frame: Where appropriate, deidentified IPD will be made accessible as noted in the data management plan filed for this study.
Access Criteria: Where appropriate, deidentified IPD will be made accessible as noted in the data management plan filed for this study.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001781-H.html